CLINICAL TRIAL: NCT05324904
Title: Intralesional Vitamin D3 Versus Intralesional Acyclovir in Treatment of Plantar Warts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, maha mostafa ali mostafa, Resident physician of Dermatology, Venereology and Andrology, kom Ombo central hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: vitamin D3, acyclovir in warts
Record Dates: First submitted 2022-03-18; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Plantar Wart
MeSH Terms: interventions — Vitamin D; Acyclovir

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Active Comparator): this group will be intralesionaly injected with vitamin D3
  Interventions: Drug: Vitamin D
- group 2 (Active Comparator): this group will be intralesionally injected with acyclovir
  Interventions: Drug: acyclovir

INTERVENTIONS:
Drug: Vitamin D — - Vitamin D
  * The aqueous solution of vitamin D3 (cholecalciferol) will be used ampoule 200,000 IU/2 ML,
  * Using a 27-gauge syringe with the bevel facing upward, a maximum of 0.6 ml (60,000 IU) of vitamin D3 solution will be slowly injected into the base of the largest plantar wart (large warts > 10 mm need multiple injections at different sites)
  * Treatment sessions will be performed at 3-week intervals for a maximum of 4 sessions
  Arms: group 1
Drug: acyclovir — -Acyclovir
  * Acyclovir vial (Zovirax® vial, 250mg, ) will be diluted with 3.5 ml saline to get approximately 70 mg /ml solution.
  * After sterilization of the skin, a 27-gauge syringe with the bevel facing upward will be inserted into the base of the largest plantar wart to slowly inject the solution
  * Treatment sessions will be performed at 2-week intervals for maximum of 5 sessions
  Arms: group 2

SUMMARY:
To evaluate and compare the efficacy and safety of intralesional acyclovir versus intralesional vitamin D3 in the treatment of plantar warts

DETAILED DESCRIPTION:
Introduction Warts are common epidermal growths caused by various strains of human papillomavirus (HPV) affecting all age groups. They have an unsightly appearance and are mostly asymptomatic but sometimes may be painful as in the case of palmoplantar warts . Plantar warts is a clinical variant that occur on sole of the foot, most frequently over pressure points .

It is estimated that 40% of population is infected with HPV, and in 7% to 12%, a wart develops . Plantar warts exhibit an annual incidence of 14% in the general population . Sixty-five percent to 78% of cutaneous warts have been shown to regress within 2 years . In persons older than 12 years, the rate of spontaneous regression significantly decreases .

Variable therapeutic options are available for treating warts, with none considered a gold standard. Primary treatments include topical salicylic acid, topical imiquimod, topical 5-fluorouracil, cryotherapy, excision, electrocautry and laser vaporization .

Vitamin D is a fat-soluble steroid prohormone that has wide range of biological actions e.g. inhibition of cellular proliferation, induction of terminal differentiation, and inhibition of angiogenesis. It also stimulates macrophages and cathelicidin production . Recently, several studies have demonstrated the efficacy of intralesional vitamin D in treatment of warts, as well as recalcitrant lesions, with clearance rates of 72.5%-90% .

Acyclovir is a synthetic purine nucleoside analogue with activity against some viruses as herpes simplex and varicella-zoster virus. Acyclovir uses viral thymidine kinase to convert to its active form, acyclovir triphosphate. Through this mechanism of utilizing viral thymidine kinase, acyclovir specifically targets viral DNA preventing its replication in the host.

Previously, few studies and case reports documented the clearance of warts, some were unresponsive to prior treatment, with both topical and oral use of acyclovir .

A recent study has evaluated the efficacy of intralesional acyclovir versus intralesional saline in treatment of warts and reported complete clearance rate of 52.6% and a partial response of 16.7% for acyclovir with a statistically significant difference from saline (0% complete clearance) .

ELIGIBILITY:
Inclusion Criteria:

* Adult participants of both sex with plantar warts will be included in the study

Exclusion Criteria:

* - Children < 12 years.
* Pregnant and lactating women.
* Receiving any treatment for warts within 1 month before the study.
* Systemic antiviral medication.
* Previous history of vitamin D or acyclovir hypersensitivity.
* Vitamin D supplementation.
* Concurrent other skin disorders.
* Immunosuppressive disorders or receiving immunosuppressive drugs.
* Receiving drugs that may alter vitamin D level including prednisone, orlistat, phenytoin and thiazide diuretics.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
complete healing rate | 12 weeks
  Main outcome variable is the complete healing rate among planter warts patients treated with intralesional vitamin D3 compared to those by Intralesional acyclovir

CONTACTS AND LOCATIONS:
Overall Officials: maha m mostafa, MD, Principal Investigator — Assuit University faculty of medicine
Locations (1):
- Assuit University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No